CLINICAL TRIAL: NCT03378063
Title: Stem Cells for Bronchopulmonary Dysplasia: a Cohort Study
Brief Title: Stem Cells for Bronchopulmonary Dysplasia
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: no stell cell accessed
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Chongqing Maternal and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: stem cell for BPD
Record Dates: First submitted 2017-12-06; First posted 2017-12-19 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2021-02

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transplantation of mesenchymal stem cell (Experimental): transplantation of mesenchymal stem cell will be given to the infants with BPD.
  Interventions: Drug: transplantation of mesenchymal stem cell
- no transplantation of mesenchymal stem cell (Active Comparator): transplantation of mesenchymal stem cell will be not given to the infants with BPD.
  Interventions: Drug: no transplantation of mesenchymal stem cell

INTERVENTIONS:
Drug: transplantation of mesenchymal stem cell — allogeneic human umbilical cord blood (hUCB)-derived mesenchymal stem cell (MSC) transplantation will be given to preterm infants
  Arms: transplantation of mesenchymal stem cell
Drug: no transplantation of mesenchymal stem cell — MSC transplantation will be not given to preterm infants
  Arms: no transplantation of mesenchymal stem cell

SUMMARY:
Very preterm infants are at high risk to develop to bronchopulmonary dysplasia (BPD) for the lack of effective measures to prevent or ameliorate this common and serious disorder. BPD remains a major cause of mortality and lifelong morbidity in preterm infants

DETAILED DESCRIPTION:
Several studies have shown that transplantation of mesenchymal stem cells (MSCs) in immunocompetent animals attenuates lung injury, such as impaired alveolarization, inflammatory response, increased apoptosis, and fibrosis. Human umbilical cord blood (hUCB) is considered a better source of MSCs because of their ready availability and greater proliferative capacity and less antigenicity than other cell types.

transplantation of hUCB-derived MSCs should be effective in treating BPD. The safety and efficacy of MSC transplantation for prevention of BPD has not been tested previously, however.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with BPD

Exclusion Criteria:

* parents' rejection

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
death | within two years
  the infant is dead due to lung disease

SECONDARY OUTCOMES:
Bayley Scales of Infant Development | 30 months after birth
  scores of Bayley Scales of Infant Development at 2 months old and 2 years old

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Daping Hospital, Research Institute of Surgery, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided